CLINICAL TRIAL: NCT01893307
Title: Phase III Randomized Trial of Intensity-Modulated Proton Beam Therapy (IMPT) Versus Intensity-Modulated Photon Therapy (IMRT) for the Treatment of Oropharyngeal Cancer of the Head and Neck
Brief Title: Intensity-Modulated Proton Beam Therapy or Intensity-Modulated Photon Therapy in Treating Patients With Stage III-IVB Oropharyngeal Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-0825; NCI-2013-01879 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0825 (Other: M D Anderson Cancer Center); R03CA188162 (NIH); R56DE025248 (NIH); U19CA021239 (NIH)
Record Dates: First submitted 2013-07-02; First posted 2013-07-09 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Stage III Oropharyngeal Squamous Cell Carcinoma AJCC v7; Stage IVA Oropharyngeal Squamous Cell Carcinoma AJCC v7; Stage IVB Oropharyngeal Squamous Cell Carcinoma AJCC v7
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy, Intensity-Modulated; Radiation; Proton Therapy; Protons

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (IMRT) (Experimental): Patients undergo IMRT QD five days a week for approximately 6.5 weeks.
  Interventions: Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Radiation: Photon Beam Radiation Therapy; Other: Quality-of-Life Assessment
- Arm II (IMPT) (Experimental): Patients undergo IMPT QD five days a week for approximately 6.5 weeks.
  Interventions: Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Radiation: Proton Beam Radiation Therapy; Other: Quality-of-Life Assessment

INTERVENTIONS:
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
  Arms: Arm I (IMRT)
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMPT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
  Arms: Arm II (IMPT)
Other: Laboratory Biomarker Analysis — Correlative studies
Radiation: Photon Beam Radiation Therapy — Undergo IMRT
  Other Names: Photon EBRT; Photon External Beam Radiotherapy; Radiation, Photon Beam
  Arms: Arm I (IMRT)
Radiation: Proton Beam Radiation Therapy — Undergo IMPT
  Other Names: PBRT; Proton; Proton EBRT; Proton External Beam Radiotherapy; Proton Radiation Therapy; Radiation, Proton Beam
  Arms: Arm II (IMPT)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase III trial studies the side effects and how well intensity-modulated proton beam therapy works and compares it to intensity-modulated photon therapy in treating patients with stage III-IVB oropharyngeal cancer. Radiation therapy uses high-energy x-rays, protons, and other types of radiation to kill tumor cells and shrink tumors. It is not yet known whether intensity-modulated proton beam therapy is more effective than intensity-modulated photon therapy in treating oropharyngeal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

To compare the progression-free survival (PFS) between concurrent chemo-radiation strategies with IMRT and IMPT following the treatment of oropharyngeal tumors.

SECONDARY OBJECTIVES:

1. To assess and compare overall survival between IMRT and IMPT along with estimating disease-related outcomes such as: [2-year progression-free survival, patterns of failure, 2-year overall survival, 2-year distant metastasis free survival, and second primary cancers]
2. To assess acute and chronic/late side effects, and to compare the rates of Grade 3-5 toxicity between IMRT and IMPT following the treatment of oropharyngeal tumors.
3. To assess Patient Reported Outcome (PRO) measures of symptoms using MD Anderson Symptom Inventory (MDASI), MD Anderson Dysphagia Inventory (MDADI), FACT-HN, Xerostomia and Health Questionnaire (EQ-5D-3L), Work status (WPAI: SHP)
4. To assess Physician Reported Toxicity using Common Terminology Criteria for Adverse Events (CTCAE)-4.0
5. To evaluate and compare Quality-Adjusted-Life-Years (QALY) between IMPT and IMRT;
6. To perform Cost-benefit economic analysis of treatment;
7. To determine whether specific molecular profiles are associated with overall or progression-free survival;
8. To investigate associations between changes in blood biomarkers, or HPV-specific cellular immune responses, or HPV ctDNA (measured at baseline and three months and at each follow-up visit for up to 10 years) with overall or progression-free survival;
9. To bank peripheral blood at time of enrollment, weeks 2, 4, and 6 during treatment and at each follow up visits for up to 10 years to explore the ability of circulating markers to predict outcome;
10. To bank head and neck tissues to explore the ability of tissue-based markers to predict outcome;
11. To bank peripheral blood and tissues for future interrogations; Finally, all additional secondary endpoints

EXPLORATORY OBJECTIVE:

I. To assess potential differences between patients on study and patients who were considered eligible for randomized, were randomized to a treatment arm, but were denied insurance coverage for the treatment arm she/he was randomized to; or may have dropped out of the study for other reasons after being randomized. These patients will compromise Group 3: consisting of patients randomized to Protons but not treated and Group 4: consisting of patients randomized to IMRT but not treated at the designated institution. Furthermore, these patients will only be followed for recurrence and survival.(Phase III)

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo IMRT once daily (QD) five days a week for approximately 6.5 weeks.

ARM II: Patients undergo IMPT QD five days a week for approximately 6.5 weeks.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 4 months for 1 year, and then every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented squamous cell carcinoma of the oropharynx (American Joint Committee on Cancer [AJCC] version [v]7 stage III-IV A,B)
* Tumor tissue (primary or cervical metastasis) available for human papilloma virus (HPV) and/or p16 (in situ hybridization [ISH], immunohistochemistry [IHC] or genotyping testing); if you do not have enough leftover tumor tissue available, you will have a tumor biopsy for tumor marker testing
* Eastern Cooperative Oncology Group (ECOG) performance status = 0, 1, or 2
* Negative pregnancy test for women of child bearing potential
* Concurrent chemotherapy
* Bilateral neck radiation

Exclusion Criteria:

* Previous radiation treatment for head and neck mucosal primary cancers within the past 5 years (i.e. oropharynx, nasopharynx, hypopharynx, larynx, and oral cavity)
* Pregnant or breast-feeding females
* Clinically significant uncontrolled major cardiac, respiratory, renal, hepatic, gastrointestinal or hematologic disease but not limited to:

  * Symptomatic congestive heart failure, unstable angina, or cardiac dysrhythmia not controlled by pacer device
  * Myocardial infarction within 3 months of registration
* Distant metastases (stage IV C, any T, any N and M1)
* Previous surgical resection or neck dissection for oropharyngeal cancer, administered with therapeutic intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2013-08-26 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of late onset grade 3+ toxicity anytime (Phase II) | Up to 2 years
  Will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The methods described by Gooley will be used to estimate the cumulative incidence of late onset grade 3+ toxicity by 2 years for each treatment arm with death as a competing risk. The methods of Fine and Gray will be used to model the cumulative incidence of late onset grade 3+ toxicity by 2 years as a function of treatment arm and other potential prognostic factors (e.g., human papillomavirus (HPV)/p16 status, use of induction chemotherapy) considering death as a competing risk. Hazard ratios for the prognostic factors from this model with 95% confidence intervals will be estimated.
Cumulative incidence of acute grade 3+ toxicity (Phase II) | Up to 2 years
  Will be graded according to the NCI CTCAE version 4.0. The methods described by Gooley will be used to estimate the cumulative incidence of late onset grade 3+ toxicity by 2 years for each treatment arm with death as a competing risk. The methods of Fine and Gray will be used to model the cumulative incidence of late onset grade 3+ toxicity by 2 years as a function of treatment arm and other potential prognostic factors (e.g., HPV/p16 status, use of induction chemotherapy) considering death as a competing risk. Hazard ratios for the prognostic factors from this model with 95% confidence intervals will be estimated.
Overall survival (OS) (Phase II) | Up to 5 years
  Stratified by treatment arm and estimated using the product limit estimator of Kaplan and Meier. Cox proportional hazards regression will be used to model OS as a function of potential prognostic factors. Hazard ratios for the prognostic factors from this model will be estimated with 95% confidence intervals.
Overall survival (Phase III) | Up to 5 years
  Will be summarized at critical time points using the method of Kaplan-Meier. Kaplan-Meier plots will be used to visualize the time-to-event information by treatment arm, and the trial will be monitored based on results from log-rank tests used to compare treatment arms. Furthermore, Cox proportional hazards regression will be used to assess the time-to-event outcomes while adjusting for covariates of interest.
Progression-free survival (Phase III) | Up to 3 years
  Will be summarized at critical time points using the method of Kaplan-Meier. Kaplan-Meier plots will be used to visualize the time-to-event information by treatment arm, and the trial will be monitored based on results from log-rank tests used to compare treatment arms. Furthermore, Cox proportional hazards regression will be used to assess the time-to-event outcomes while adjusting for covariates of interest.

SECONDARY OUTCOMES:
Quality of life (QoL) (Phase II and III) | Up to 5 years
  QoL assessments will be summarized using the mean score and standard deviation for each time point of interest. Mean response trajectories will be plotted over the time horizon for each QoL instrument administered to patients in order to explore differences between treatment arms along with other patient characteristics of interest. Other analyses such as area under the curve and linear mixed models will be used to make statistical comparisons between treatment arms while adjusting for covariates of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Frank, Principal Investigator — M.D. Anderson Cancer Center
Locations (22):
- United States (22):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Miami Cancer Institute, Miami, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Willis-Knighton Medical and Cancer Center, Shreveport, Louisiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - New York Proton Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson in The Woodlands, Conroe, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

REFERENCES:
- [Derived] Frank SJ, Busse PM, Lee JJ, Rosenthal DI, Hernandez M, Swanson DM, Garden AS, Gunn GB, Patel SH, Snider JW, Ma DJ, Molitoris JK, Lee NY, Parvathaneni U, McDonald MW, Kalman NS, Lin A, Mohammed N, Henson C, Hyde C, Bajaj GK, Katz SR, Dagan R, Morrison WH, Reddy JP, Fuller CD, Shah SJ, Phan J, Chronowski GM, Mayo L, Sturgis EM, Ferrarotto R, Zhu XR, Zhang X, Wang L, Hutcheson KA, El-Naggar AK, Moreno AC, Lee A, Spiotto MT, Gross ND, Lai SY, Liao JJ, Paly J, Liao Z, Foote RL; University of Texas MD Anderson Cancer Center Clinical Trial Consortium. Proton versus photon radiotherapy for patients with oropharyngeal cancer in the USA: a multicentre, randomised, open-label, non-inferiority phase 3 trial. Lancet. 2026 Jan 10;407(10524):174-184. doi: 10.1016/S0140-6736(25)01962-2. Epub 2025 Dec 11. PMID 41391462
- [Derived] Moreno A, Sahli AJ, Johnson F, Sun X, Barbon C, Rinsurongkawong W, Song W, Luciani FM, Liang H, Li J, Liu W, Lee JJ, Frank SJ, Lai S, Fuller C, Hutcheson K; P01 MD Anderson Oropharynx Cancer Program. Stiefel MD Anderson OroPharynx cancer (MDA-OPC) cohort: a single-institution, prospective longitudinal outcomes study. BMJ Open. 2025 Nov 24;15(11):e106845. doi: 10.1136/bmjopen-2025-106845. PMID 41290309
- [Derived] Gunn GB, Blanchard P, Garden AS, Zhu XR, Fuller CD, Mohamed AS, Morrison WH, Phan J, Beadle BM, Skinner HD, Sturgis EM, Kies MS, Hutcheson KA, Rosenthal DI, Mohan R, Gillin MT, Frank SJ. Clinical Outcomes and Patterns of Disease Recurrence After Intensity Modulated Proton Therapy for Oropharyngeal Squamous Carcinoma. Int J Radiat Oncol Biol Phys. 2016 May 1;95(1):360-367. doi: 10.1016/j.ijrobp.2016.02.021. Epub 2016 Feb 12. PMID 27084653
- See also: M D Anderson Cancer Center website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2025-01-22): https://cdn.clinicaltrials.gov/large-docs/07/NCT01893307/ICF_000.pdf